CLINICAL TRIAL: NCT00811330
Title: Interest of Statin in Surgical Aortic Stenosis: From Myocardial Preconditioning to Ventricular Reverse Remodeling.
Brief Title: Effects of High Dose Atorvastatin in Patients With Surgical Aortic Stenosis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3963
Record Dates: First submitted 2008-12-17; First posted 2008-12-19 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-06

CONDITIONS: Aortic Valve Stenosis; Ventricular Hypertrophy
Keywords: Left ventricular hypertrophy; Aortic valve stenosis; Aortic valve replacement; Cardiopulmonary bypass; Statins; Myocardial preconditioning; Left ventricular reverse remodeling
MeSH Terms: conditions — Aortic Valve Stenosis; Hypertrophy, Left Ventricular | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: Atorvastatin 80 mg. (Experimental): Atorvastatin 80 mg PO every day for one year. The treatment will start 4 weeks before aortic valve replacement.
  Interventions: Drug: Atorvastatin 80 mg
- 2: No Atrovastatine (No Intervention)

INTERVENTIONS:
Drug: Atorvastatin 80 mg — Atorvastatin 80 mg PO every day for one year. The treatment will start 4 weeks before aortic valve replacement.
  Arms: 1: Atorvastatin 80 mg.

SUMMARY:
The purpose of the study is to see if statin therapy will optimize myocardial response to cardiopulmonary bypass during aortic valve replacement (AVR) for aortic valve stenosis (AVS) (Phase I) and optimize left ventricular reverse remodeling following AVR (Phase II). Preliminary evidence indicates that perioperative statin therapy reduce mortality and morbidity following cardiac surgery. Pleiotropic effects of statins may induce myocardial preconditioning and optimize myocardial and systemic responses to cardiopulmonary bypass during AVR. Furthermore statin therapy after AVR may contribute to an optimal left ventricular reverse remodeling.

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 70 years and < 80 years
* Severe aortic valve stenosis
* Indication for aortic valve replacement by bioprothesis
* Ejection fraction > or = 50%
* Without treatment with statin- No renal failure
* Informed consent signed

Exclusion Criteria:

* Ischemic heart disaese
* Concomitant surgery to aortic valve replacement
* Emergency surgery- Known intolerance for statin
* Pregnant woman

Ages: 70 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-12; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
♦ Phase I: To study changes on inflammatory markers after aortic valve replacement. ♦ Phase II: To study changes in left ventricular mass at the end of the study (12 months). | 1 year

SECONDARY OUTCOMES:
Phase I: To study changes on mitochondrial function, reactive oxygen species, and perioperative systolic and diastolic functions. Phase II: To study changes on clinical status, systolic and diastolic functions during the one-year follow-up. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Michel KINDO, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service de Chirurgie Cardio-VasculaireHôpital Civil, Strasbourg, France